CLINICAL TRIAL: NCT03087747
Title: Percutaneous Drainage in a Setting of Acute Cholecystitis Severity Grade III and Correlation With Clinical Outcomes
Brief Title: Percutaneous Transhepatic Cholangiography (PTHC) in Acute Cholecystitis and Clinical Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: poor accrual
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Marija Cavar, MD, University of Split, School of Medicine
Other Study IDs: AChol
Record Dates: First submitted 2017-03-07; First posted 2017-03-22 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Cholecystitis, Acute; Elderly Infection; Drain Abscess
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients older than 80 yr. Clinical parameters after percutaneous transhepatic cholangiography (PTHC).
  Interventions: Procedure: Percutaneous cholecystostomy
- Group 2: Patients younger than 80 yr. Clinical parameters after percutaneous transhepatic cholangiography (PTHC).
  Interventions: Procedure: Percutaneous cholecystostomy

INTERVENTIONS:
Procedure: Percutaneous cholecystostomy — Placement of drainage catheter into gallbladder lumen in order to evacuate inflamed content.

SUMMARY:
In a setting of acute cholecystitis (AC) one of the treatment option is percutaneous transhepatic cholangiography (PTHC) drainage. The goal of current study is to evaluate some radiology aspects and correlate with clinical patient outcomes in patients with acute cholecystitis severity grade III (presented as acute cholecystitis with organ dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* clinical markers of acute cholecystitis
* diagnosis confirmed with some imaging technique: computed tomography (CT), ultrasound (US).

Exclusion Criteria:

* clinical diagnosis was not confirmed with imaging.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute cholecystitis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein (CRP) | Up to 8 weeks.
  C-reactive protein (CRP) is a protein found in blood plasma, whose levels rise in response to inflammation.

SECONDARY OUTCOMES:
Drainage duration (expressed in days) | Up to 16 weeks.
  The drain which is placed in gallbladder during Percutaneous transhepatic cholangiography (PTHC) remains there until resolving clinical parameters of acute cholecystitis.
White blood cells (WBCs) count | Up to 8 weeks.
  White blood cells (WBCs) are the cells of the immune system. During inflammation White blood cell level rise.

CONTACTS AND LOCATIONS:
Overall Officials: Liana Cambj Sapunar, Professor, Study Director — University Hospital of Split
Locations (1):
- University of Split, School of Medicine, Split, Croatia